CLINICAL TRIAL: NCT06886529
Title: Early PACT Involvement in Cardiology Patients Using Machine Learning
Brief Title: PACT Involvement in Cardiology Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Lillian Sung, Chief Clinical Data Scientist, Paediatric Oncologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 3433
Record Dates: First submitted 2025-03-13; First posted 2025-03-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Machine Learning; Cardiovascular Outcome; Pediatric Palliative Care; Pediatric Cardiology
Keywords: quality of life; cardiovascular outcomes; machine learning; prediction models; pediatric

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ML model (Experimental): Cardiac patients identified by an ML model for having the highest risk of serious cardiac outcomes.
  Interventions: Other: ML-based intervention

INTERVENTIONS:
Other: ML-based intervention — ML model predicting a serious cardiac event in cardiac patients, defined as VAD procedure, being wait listed for heart transplant or death within the next three months.

SUMMARY:
The goal of this trial is to determine the effectiveness of a machine-learning (ML) model predicting a serious cardiac event within the next three months, when compared pre- versus post-deployment, in pediatric cardiac inpatients. The main questions it aims to answer are whether deployment of the ML model:

1. Increases PACT consultation within the next three months among admissions without PACT involvement in the previous 100 days
2. Increases PACT consultation or visit within the next three months among those who experience a serious cardiac event during this period
3. Decreases time to PACT consultation or visit among those seen by PACT during this period
4. Decreases the incidence of death in the intensive care unit (ICU)
5. Increases documentation of goals of care

High-risk cardiology patients will be identified by an ML model each morning. If the patient has been seen by the PACT team within the past year, the update will go to the PACT team members. If the patient hasn't been seen by the PACT team, the email will be sent to the cardiology physician in charge of the patient. This physician will decide whether a PACT consultation is necessary based on their clinical judgment. If so, a referral will be made using the usual process. Outcomes of the identified patients will be compared pre- and post-deployment.

DETAILED DESCRIPTION:
At The Hospital for Sick Children (SickKids), the collaboration between cardiology and palliative care is much stronger than other centers, with routine involvement in patients being considered for heart transplant. Despite this, earlier involvement of palliative care would be advantageous. Our cardiology co-investigators identified patients who would benefit from earlier palliative care team involvement as those receiving advanced heart therapies (defined as ventricular assist device (VAD) and being wait listed for heart transplant) and those who die. The study team created a clinical deployment environment named SickKids Enterprise-wide Data in Azure Repository (SEDAR). [1] SEDAR is a modular and robust approach to deliver foundational data that is re-usable across multiple ML projects. It offers validated EHR data in a standardized and curated schema. ML is a promising approach to identify cardiac patients at the highest risk of these serious cardiac outcomes who may benefit from earlier palliative care team involvement. To assess the effectiveness of this approach, patient outcomes will be compared pre- and post-deployment of the ML model. The pre-period will include patients admitted for a 12-month period before deployment (starting 15 months prior to deployment). The post-period will include patients admitted for a 12-month period following deployment starting 3 months post-deployment start.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric inpatients admitted to cardiology

Exclusion Criteria:

* Expected to be discharged prior to midnight on the day of admission

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2027-06-28 (Estimated); Study Completion 2027-06-28 (Estimated)

PRIMARY OUTCOMES:
Proportion of admissions with PACT consultation within the next three months among admissions without PACT involvement in the previous 100 days | Time of enrolment to 3 months
  The primary outcome will be the proportion of admissions with PACT consultation within the next three months among admissions without PACT involvement in the previous 100 days. This variable will be measured using SEDAR.

SECONDARY OUTCOMES:
PACT consultation or visit within the next three months among those with a positive model prediction | Time of enrolment to 3 months
  PACT consultation or visit within the next three months among those with a positive model prediction will be measured using SEDAR.
Time to PACT consultation or visit among those seen by PACT | Time of enrolment to 3 months
  Time to PACT consultation or visit among those seen by PACT will be measured using SEDAR.
Death in the ICU | Time of enrolment to 3 months
  Death in the ICU will be measured using SEDAR.
Documentation of goals of care | Time of enrolment to 3 months
  Goals of care will be abstracted via chart review.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Sung, MD, PhD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patel P, Robinson PD, Phillips R, Baggott C, Devine K, Gibson P, Guilcher GMT, Holdsworth MT, Neumann E, Orsey AD, Spinelli D, Thackray J, van de Wetering M, Cabral S, Sung L, Dupuis LL. Treatment of breakthrough and prevention of refractory chemotherapy-induced nausea and vomiting in pediatric cancer patients: Clinical practice guideline update. Pediatr Blood Cancer. 2023 Aug;70(8):e30395. doi: 10.1002/pbc.30395. Epub 2023 May 13. PMID 37178438